CLINICAL TRIAL: NCT01019057
Title: A Prospective, Non-randomized, Multi-Center Evaluation of Interlaminar Lumbar Instrumented (ILIF™)
Brief Title: An Evaluation of Interlaminar Lumbar Instrumented (ILIF™)
Acronym: ILIF
Status: Completed | Type: Observational
Sponsor: NuVasive (Industry)
Responsible Party: Sponsor
Organization: Globus Medical Inc (Industry)
Other Study IDs: NUVA.IL.0901
Record Dates: First submitted 2009-11-23; First posted 2009-11-25 (Estimated); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Degenerative Disc Disease
Keywords: DDD; decompression; spinous process plate
MeSH Terms: conditions — Intervertebral Disc Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ILIF — Interlaminar lumbar instrumented fusion (ILIF™) is a compound surgical solution to spinal stenosis, combining direct neural decompression with an allograft interspinous spacer (ExtenSure® H2) to maintain the segmental distraction, and a spinous process fixation plate (Affix™) to maintain stability for eventual segmental fusion.

SUMMARY:
Patients diagnosed with single-level degenerative disc disease (DDD) of the lumbar spine undergo a posterior decompression followed by a fusion complete with a spinous process plate, graft, and a biologic.

DETAILED DESCRIPTION:
Interlaminar lumbar instrumented fusion (ILIF™) is a compound surgical solution to spinal stenosis, combining direct neural decompression with an allograft interspinous spacer (ExtenSure® H2) to maintain the segmental distraction, and a spinous process fixation plate (Affix™) to maintain stability for eventual segmental fusion. Because this compound solution requires only a midline incision rather than the far lateral exposure necessary in posterolateral fusion with pedicle screws, it is less invasive to the patient, and therefore should result in less postoperative pain and disability, broadening the applicability of the procedure to even those advanced in age or with existing comorbidities. Subjects will be followed for 24 months following surgery to determine the changes in ODI scores from preoperative to baseline assessments. This data will be compared to published data on similar procedures.

ELIGIBILITY:
Inclusion Criteria:

* Patient is over 40 years of age;
* Patient is diagnosed with single-level lumbar degenerative disc disease between L1-L2 and L4-L5 with evidence of disc collapse and symptomatic claudication with or without back pain and requires surgical intervention;
* Patient is unresponsive to conservative treatment greater than or equal to six month 6 months, or exhibits progressive neurological symptoms in the face of conservative treatment;
* Patient is willing and able to comply with the requirements defined in the protocol for the duration of the study;
* Patient has signed and dated Informed Consent.

Exclusion Criteria:

* Patients with lumbar pathologies requiring surgical treatment at more than one level;
* Patients with spondylolisthesis > grade 1;
* Patients with lytic spondylolisthesis or a defect of the pars interarticularis;
* Patients with prior lumbar surgery at or adjacent to the operative level;
* Patients with spinal metastases or active spinal tumor malignancy;
* Progressive neuromuscular disease, e.g., muscular dystrophy, multiple sclerosis;
* Present chronic steroid use;
* Patients with rheumatoid arthritis or other autoimmune disease;
* Patients who are pregnant or interested in becoming pregnant within the follow-up period of the study;
* Patients with a history of substance abuse;
* Patients involved in active spinal litigation;
* Patients receiving workman's compensation for spinal conditions;
* Patients who are mentally incompetent;
* Patients who are incarcerated;
* Patients who are unwilling or unable to comply with the follow-up protocol schedule of visits and assessments.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study populuation will be comprised of 50 patients across different cities in the United States.
Sampling Method: Non-Probability Sample
Enrollment: 77 (Actual)
Dates: Start 2009-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
The change in Oswestry Disability Index scores at 24 months compared to baseline. | preoperative to 24 months follow-up

SECONDARY OUTCOMES:
The change in subject self-reported pain ratings (VAS scores) at 24 months compared to baseline | pre-op to 24 months follow-up
The change in Zurich Claudication Questionnaire scores at 24 months compared to baseline | pre-op to 24 months follow-up
The rate of surgical and/or postoperative complications attributable to ILIF™ requiring secondary surgical intervention | pre-op to 24 months follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Bae, M.D, Principal Investigator — The Spine Institute in Los Angeles, CA
Locations (8):
- United States (8):
  - Desert Institute for Spine Care, Surgical Specialty Hospital of Arizona, Phoenix, Arizona
  - The Spine Institute, St. John's Health Center, Santa Monica, California
  - North Florida Regional Medical Center, Gainesville, Florida
  - Lovelace Medical Center, Albuquerque, New Mexico
  - Coastal Orthopaedic Associates PA, Conway, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Center for Neurological Disorders, Texas Health Harris Methodist Fort Worth, Fort Worth, Texas
  - Neurosurgical Specialists, DePaul Medical Center, Norfolk, Virginia

REFERENCES:
- See also: Related Info — http://www.nuvasive.com